CLINICAL TRIAL: NCT05265767
Title: Gene Therapy for Hemophilia A With a High Expression Factor VIII Transgene in Autologous Hematopoietic Stem Cells
Brief Title: Hematopoietic Stem Cell Transplantation Gene Therapy for Treatment of Severe Hemophilia A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Christian Medical College, Vellore, India (Other)
Collaborators: Dr. H. Trent Spencer, Professor, Emory University of Medicine, Atlanta Ga, 30322 (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSCR-CMC/FVIII LVGT/2018
Record Dates: First submitted 2022-02-16; First posted 2022-03-04 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Intervention Model Description: Patients with Severe haemophilia A
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Autologous HSCT CD68-ET3-LV gene therapy (Experimental): Autologous gene modified peripheral blood stem cell transplantation for patients with severe hemophilia A (FVIII <1%).
  Interventions: Biological: Auto CD34+PBSC transduced with a lentiviral vector encoding a novel coagulation factor VIII transgene

INTERVENTIONS:
Biological: Auto CD34+PBSC transduced with a lentiviral vector encoding a novel coagulation factor VIII transgene — Auto CD34+PBSC transduced with a lentiviral vector encoding a novel coagulation factor VIII transgene administered by IV infusion following conditioning regimen.

SUMMARY:
Factor VIII (FVIII) is a large plasma glycoprotein that participates in blood coagulation. Loss of circulating FVIII activity due to mutations within the F8 gene results in the X-linked, recessive bleeding disorder hemophilia A. The clinical presentation ranges from a mild to severe bleeding phenotype that correlates with the patient's residual plasma FVIII activity level.

Current state of the art treatment entails frequent infusion of FVIII protein. However, several limitations remain to treating hemophilia A, which are 1) access to FVIII-replacement products (currently <30% of the world population is treated adequately, access is highly restricted in India), 2) high burden of compliance with treatment protocols particularly in children 3) the expense of FVIII-replacement products, 4) the development of humoral anti-FVIII immune responses that block FVIII activity and limit treatment efficacy and 5) morbidity due to crippling musculoskeletal disease when inadequately treated. Several newer hemostasis agents are being developed but like the recombinant Clotting Factor Concentrate (CFC) from the 1990s, these are also not likely to be made available in India for many years. Currently, the only cure for hemophilia A is orthotopic liver transplantation.

DETAILED DESCRIPTION:
Eligible subjects will undergo (Cluster of Differentiation) CD34+ hematopoietic stem cell collection. These cells will be transduced ex vivo with (Cluster of Differentiation) CD68-ET3 lentiviral vector and subsequently, following a conditioning regimen, the transduced cells will be infused to patients. After completion of study treatment, patients are followed up periodically for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent for the protocol approved by the Institutional Review Board.
* Male subjects who are ≥18 years of age and < 45 years of age.
* Diagnosis of severe hemophilia A (<1 IU/dl factor VIII activity).
* Documented history of more than 100 exposures of factor VIII treatment.
* Average of at least 3 bleeds requiring treatment per year over the prior three years, at least 3 bleeds per year during the 3 years preceding the initiation of prophylaxis, or evidence of joint damage (knee, elbow or ankle) on physical or radiographic examination thought to be related to hemophilia.
* Performance status (Karnofsky score) of at least 70.
* Willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

* History of spontaneous central nervous system bleeding within the last 5 years.
* Significant organ dysfunction which could interfere with outcome of therapy such as: -
* Cardiac: There should be no evidence of significant cardiac dysfunction (resting left ventricular ejection fraction of < 50%) and no cardiomegaly. There should not be uncontrollable hypertension.
* Renal: Glomerular Filtration Rate (GFR) < 60 ml/min/1.73m2 as calculated using the Cockcroft-Gault equation.
* Hepatic: There should be no evidence of hepatic dysfunction which is defined as a serum bilirubin of > 1.5 mg/dl and Aspartate Amino Transferase (AST) / Alanine Amino Transferase (ALT) > 3X the upper limit of normal,
* Hematologic: Absolute neutrophil counts (ANC) < 1000/mm3 and platelets counts < 150,000/μL.
* Pulmonary function with a corrected Diffusing Capacity of lung for Carbon Monoxide (DLCO) of < 50% predicted
* History of a FVIII inhibitor (>0.6 Bethesda Units/ml) including at least 2 measurements over the preceding 5 years or any single titer >5 Bethesda Units (BU) /ml.
* Previous stem cell transplant.
* HIV positive.
* Evidence of hepatitis B active infection or chronic carrier
* Evidence of chronic hepatitis C infection. Absence of chronic infection will be documented with at least 2 negative viral loads at least 6 months apart.
* Diagnosis of a bleeding disorder other than hemophilia A
* Use of medication(s) that can affect hemostasis (e.g. aspirin and non- cyclooxygenase (COX-2) selective non-steroid anti-inflammatory drugs).
* History of cancer or familial cancer syndromes
* Any condition in the opinion of the principle investigator that will negatively impact the subject's ability to safely undergo an autologous stem cell transplant.
* Any reason in the opinion of the principle investigator that will negatively impact the subject's ability to complete the clinical trial per the trial protocol.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Hemophilia A is an inherited X-linked recessive genetic pattern, so males are commonly affected
Enrollment: 6 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Number of study participants experiencing serious adverse events (SAEs) following treatment through 12 weeks. | Percentage of patients experiencing SAEs following 12 weeks of treatment
  As assessed by physical examination, vital signs, clinical labs, and FVIII inhibitor levels (Bethesda assay). Serious adverse event (SAE) is an AE resulting in any of the following outcomes: death; Life-threatening event; Required or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly.
Severity of serious adverse events following administration of CD68-ET3-LV CD34+ as assessed by NCI Common Toxicity Criteria for Adverse Events (CTCAE) Version 5.0. | Assessement of severity of SAE through 12 weeks after treatment
  Serious adverse events severity assessment
Duration of the serious adverse events following administration of CD68-ET3-LV CD34+. | Assessment of duration of SAEs after 12 weeks of treatment
  As assessed by stop and end dates of the SAEs

SECONDARY OUTCOMES:
Time to absolute neutrophil count (ANC) recovery. | Measurement of ANC upto 5 years
  Time to ANC recovery (the first day a neutrophil count is >0.5 x 109/L (>500/µL) on three consecutive days) following busulfan/ anti-thymocyte globulin conditioning and infusion of autologous CD34+ hematopoietic stem and progenitor cells (HSPC) transduced with CD68-ET3-LV.
Time to platelet recovery | Measured of platelet recovery upto 5 years
  Time to platelet recovery (the first day a platelet count is > 50,000/µL on three consecutive days without platelet transfusions during the prior 7 days) following infusion of autologous CD34+ cells transduced with CD68-ET3-LV.
Anti-human factor VIII inhibitor titer | Measured of FVIII inhibitor titer upto 5 years
  Assessed via Bethesda assay
Immune response to ET3 as measured by modified Bethesda assay incorporating ET3i spiked into FVIII-deficient plasma | Measured of Immune response to ET3 for up to 5 years
  Immune response to ET3
Vector copy number of circulating genetically modified cells as determined by real time Polymerase Chain Reaction (PCR) | Measured of Vector copy number by PCR upto 5 years
  Vector copy number determined via real time PCR
To evaluate FVIII activity after Autologous Hematopoietic Stem Cell Transplantation (HSCT) with CD68ET3-LV transduced CD34+ cells through measurement of plasma FVIII activity levels. | Measurement of FVIII activity (assay) upto 5 years
  Evaluate FVIII activity
To evaluate the impact of autologous HSCT with CD68ET3-LV transduced CD34+ cells on bleeding phenotype as measured by frequency of bleeding episodes and clotting factor concentrate (CFC) usage. | Measured of frequency of bleeding episodes and CFC usage upto 5 years
  Evaluate the impact of autologous HSCT with CD68ET3-LV transduced CD34+ cells
To evaluate the relationship between FVIII activity level and engraftment of CD68ET3-LV modified cells. | Evaluation of relationship between FVIII activity and engraftment upto 5 years
  Evaluate correlation between FVIII activity in % level and engraftment of ANC measured in per cubic milliliter (cumm) Platelets values in per cumm

OTHER OUTCOMES:
Annualized bleed rate (ABR) assessed by number of bleeding episodes and in comparison to before gene therapy. | Assessement of Annualized bleeding rate (ABR) through long term follow-up for up to 15 years
  To evaluate the impact of autologous HSCT with CD68-ET3-LV CD34+ on annualized bleed rate.

CONTACTS AND LOCATIONS:
Overall Officials: Alok Srivastava, MD, Principal Investigator — Christian Medical College, Vellore, India
Locations (1):
- Christian Medical College Vellore Ranipet Campus, Vellore, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Srivastava A, Abraham A, Aboobacker F, Singh G, Geevar T, Kulkarni U, Selvarajan S, Korula A, Dave RG, Shankar M, Singh AS, Jeba A, Kumaar N, Benjamin C, Lakshmi KM, Srivastava VM, Shaji RV, Nair SC, Brown HC, Denning G, Lollar P, Doering CB, Spencer T. Lentiviral Gene Therapy with CD34+ Hematopoietic Cells for Hemophilia A. N Engl J Med. 2025 Jan 30;392(5):450-457. doi: 10.1056/NEJMoa2410597. Epub 2024 Dec 9. PMID 39655790